CLINICAL TRIAL: NCT02455284
Title: In Vivo and ex Vivo Validation of MR Tractography of Brain White Matter Tracts - FIBRATLAS II-III
Acronym: FIBRATLAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ANR 14 - CD / FIBRATLAS
Record Dates: First submitted 2015-05-12; First posted 2015-05-27 (Estimated); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Neurological Diseases
Keywords: MRI; Tractography; white; physiology; analysis; matter; tracts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy subjects (Experimental): MRI and neuropsychological evaluation
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — In vivo MRI with B0 cartography, FLAIR, 3D T1 anatomic images, DWI, and Tractography from DWI images

SUMMARY:
White matter tracts connect cortical areas to other parts of the cortex, to basal ganglia and to the brain stem and spinal cord. These tracts form the internal part of the brain and transmit the nervous impulses. Changes in brain white matter may serve as biomarkers for numerous neurological diseases.

Diffusion Weighted Imaging (DWI) is a non-invasive MRI (Magnetic Resonance Imaging) technique providing information on white matter tracts (tractography) by studying water diffusion. Since it is based on complex mathematical models that only indirectly evaluates the underlying anatomy, tractography need to be validated before being used for research and clinical purposes. Several validation techniques were previously proposed, none of them being fully convincing in human.

ELIGIBILITY:
Inclusion Criteria:

* Prior enrollment in a body donation program
* Age ≥ 82 years
* Absence of major cognitive impairment as demonstrated by independent living skills in 4 fields evaluated by the IADL (4 items) (Lawton and Brody, 1969)
* Distance to one of the participating laboratories ≤ 120km
* Able to remain supine in the MR scanner for acquisition duration (60 min),
* Affiliation to Social Security
* Informed and written consent

Non Inclusion Criteria:

* Past or present Neurological or Neurosurgical diseases (excluding trauma or degenerative spinal lesions)
* Uncontrolled: High blood pressure, diabetes (types I or II), or dyslipemia
* Contraindications to MRI
* Contraindication to body donation

Exclusion criteria

* Diagnosis on MRI of brain lesions, excepted common age-related changes

Min Age: 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 134 (Actual)
Dates: Start 2015-10; Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Reconstructions of the fiber tracts | 5.5 years
  similarity indices, such as modified Haussdorf distance, measured on MRI images

SECONDARY OUTCOMES:
Number of subjects included in the database | 5.5 years
  Number of subjects included in the database
Scores at neuropsychological evaluation | 5.5 years
  Scores at neuropsychological evaluation
In vivo MRI measures obtained from DWI | 5.5 years
  In vivo MRI measures obtained from DWI

CONTACTS AND LOCATIONS:
Overall Officials: Christophe DESTRIEUX, PhD, Principal Investigator — University Hospital of Tours
Locations (7):
- France (7):
  - University Hospital of Amiens, Amiens
  - University Hospital of Angers, Angers
  - University Hospital of Brest, Brest
  - Hospital of Charpennes - Lyon, Lyon
  - University Hospital of Nancy, Nancy
  - University Hospital of Rennes, Rennes
  - University Hospital of Tours, Tours

REFERENCES:
- [Result] Sizaret E, Brachet M, Launay A, Destrieux C, Zemmoura I, Angel L; FIBRATLAS Consortium. Norms for neuropsychological tests in cognitively healthy French oldest old adults. J Int Neuropsychol Soc. 2024 Nov;30(9):841-855. doi: 10.1017/S1355617724000390. Epub 2024 Sep 18. PMID 39291410